CLINICAL TRIAL: NCT04757714
Title: Thoracic Kyphosis and Osteoporosis: Study of Their Relationship With Respiratory Functions in Chronic Obstructive Pulmonary Disease.
Acronym: CYPHOS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The site is no more able to conduct the study
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHRO-2020-05
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: COPD; Osteoporosis; Kyphosis
Keywords: osteoporosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Osteoporosis; Kyphosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD Patients (Other): Patients agreeing to participate in the study and meeting the inclusion and non-inclusion criteria will have:
  * The high-resolution peripheral scanner (HRpQCT) of the tibia and radius
  * a low-dose imaging system exploration of their thoraco-lumbar spine (EOS system)
  * to complete:
    * a physical activity questionnaire (PHAS instrument)
    * a COPD quality of life questionnaire (St George Hospital)
  * A search for sarcopenia by studying the strength of the grip (dynamometer)
  Interventions: Procedure: The high-resolution peripheral scanner (HRpQCT) of the tibia and radius; Procedure: a low-dose imaging system exploration of their thoraco-lumbar spine (EOS system); Other: Questionnaires; Other: A search for sarcopenia by studying the strength of the grip (dynamometer)

INTERVENTIONS:
Procedure: The high-resolution peripheral scanner (HRpQCT) of the tibia and radius — The high-resolution peripheral scanner (HRpQCT) of the tibia and radius
Procedure: a low-dose imaging system exploration of their thoraco-lumbar spine (EOS system) — a low-dose imaging system exploration of their thoraco-lumbar spine (EOS system)
Other: Questionnaires — * a physical activity questionnaire (PHAS instrument)
  * a COPD quality of life questionnaire (St George Hospital)
Other: A search for sarcopenia by studying the strength of the grip (dynamometer) — A search for sarcopenia by studying the strength of the grip (dynamometer)

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a condition characterized by a progressive and incompletely reversible limitation of airborne gas flow . The association of co-morbidities with COPD and acute flare-ups of respiratory failure contribute to the overall severity of this disease. The prevalence of COPD is high, affecting up to 10% of people over the age of 40 years and causing high morbidity and mortality rates. While COPD is a disease primarily affecting the lungs, it is associated with many extra-pulmonary conditions including sleep apnea, depression, anemia, chronic kidney failure, wasting, cardiovascular disease, skeletal muscle weakness and osteoporosis (OP).

DETAILED DESCRIPTION:
Osteoporosis, characterized by bone quality disorders and low bone mineral density (BMD) leading to a high risk of fractures, is common in COPD patients. For example, studies have reported OP rates ranging from 9% to 69% in COPD patients. The explanatory factors for this low BMD are clearly multiple, involving to varying degrees of importance, vitamin D deficiency, depression, sedentary lifestyle, smoking, corticosteroids, low lean body mass and body mass index, chronic inflammation, low nutritional status, chronic hypoxia and hypercapnia. This is why patients with COPD have a high prevalence of fractures, particularly vertebral fractures (VF) ranging from 30 to 63% depending on the studies. In these patients the existence of thoracic VF is of crucial importance, as each VF is associated with a 9% decrease in the forced vital capacity of COPD patients.

For these reasons the latest HAS recommendations for COPD management indicate that the risk of osteoporosis should be systematically investigated and treated (HAS, 2014).

However, the relationship between densitometric variations and the presence of thoracic VF and the prognosis and severity of the disease is not yet very clear, as studies of these relationships have produced mixed results.

On the other hand, it is well established that patients with a recent diagnosis of COPD have a high prevalence of densitometric OPs and fractures.

Thoracic kyphosis is one of the determinants of the incidence of vertebral fractures. Increased thoracic kyphosis is associated with decreased physical capacity, increased risk of falls and abnormal respiratory function.

In addition, measurement of thoracic kyphosis was previously carried out either indirectly using point coordinates recorded in a database (patients were assessed in the supine position) or more directly using a ruler applied against the back.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman age > 40
* FEV1/CVF ratio < 0.7 as defined by the Global Initiative for Chronic Obstruction Lung Disease (GOLD).
* Moderate to severe COPD as defined by GOLD (grade C and D)

Exclusion Criteria:

* Presence of metal or plastic parts in the field of examination
* Pregnancy
* Patients who are not affiliated with or do not benefit from a social security system
* Person under guardianship or curatorship

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The thoracic kyphosis index | Day 0
  The kyphosis index will be used to assess thoracic kyphosis at the beginning of the study. This index is a percentage.
Forced vital capacity | Day 0

SECONDARY OUTCOMES:
Presence of densitometric osteoporosis | Day 0
Presence of intermediate bone density | Day 0
Percentage of maximum expiratory volume per second (FEV1), percentage predicted value | Day 0
predicted value FEV1/Forced Vital Capacity | Day 0
Quality of life score (St George Hospital questionnaire) | Day 0
Severity index of Osteoporosis | Day 0
  raw BMD values
Severity index of Osteoporosis | Day 0
  FRAX score
Severity index of Osteoporosis | Day 0
  number of VFs
Chronic Obstructive Pulmonary Disease (COPD) severity index | Day 0
  maximum expiratory volume per second (FEV1)
Chronic Obstructive Pulmonary Disease (COPD) severity index | Day 0
  severity stage by the Global Initiative for Chronic Obstruction Lung Disease (GOLD)
Chronic Obstructive Pulmonary Disease (COPD) severity index | Day 0
  prognosis stage according to BODE index
Parameters measured by HRpQCT | Day 0
  volume density and microarchitecture
Densitometric osteoporosis status | Day 0
  The status will be determine between: Osteoporosis , intermediate bone density and normal

CONTACTS AND LOCATIONS:
Overall Officials: Eric LESPESSSAILLES, Ph.D., Principal Investigator — CHR ORLEANS
Locations (1):
- CHR d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Cielen N, Maes K, Gayan-Ramirez G. Musculoskeletal disorders in chronic obstructive pulmonary disease. Biomed Res Int. 2014;2014:965764. doi: 10.1155/2014/965764. Epub 2014 Mar 25. PMID 24783225
- [Background] Decramer M, Janssens W, Miravitlles M. Chronic obstructive pulmonary disease. Lancet. 2012 Apr 7;379(9823):1341-51. doi: 10.1016/S0140-6736(11)60968-9. Epub 2012 Feb 6. PMID 22314182
- [Background] Eagan TM, Aukrust P, Ueland T, Hardie JA, Johannessen A, Mollnes TE, Damas JK, Bakke PS, Wagner PD. Body composition and plasma levels of inflammatory biomarkers in COPD. Eur Respir J. 2010 Nov;36(5):1027-33. doi: 10.1183/09031936.00194209. Epub 2010 Apr 22. PMID 20413541
- [Background] Ekblom O, Ekblom-Bak E, Bolam KA, Ekblom B, Schmidt C, Soderberg S, Bergstrom G, Borjesson M. Concurrent and predictive validity of physical activity measurement items commonly used in clinical settings--data from SCAPIS pilot study. BMC Public Health. 2015 Sep 28;15:978. doi: 10.1186/s12889-015-2316-y. PMID 26415512